CLINICAL TRIAL: NCT07227376
Title: Data Collection Using Eko Digital Devices in a Clinical Setting
Status: Recruiting | Type: Observational
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022.5 V10.0
Record Dates: First submitted 2025-10-24; First posted 2025-11-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Lung Diseases
Keywords: lung sounds; adventitious lung sounds; abnormal lung sounds
MeSH Terms: conditions — Lung Diseases; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Eko digital stethoscopes — Use of the Eko CORE 500 digital stethoscope and 3M Littmann CORE Digital Stethoscope to listen for and record lung sounds.

SUMMARY:
The purpose of this research is to prospectively train and validate an artificial intelligence machine learning (ML) algorithm to detect the presence of adventitious lung sounds in adults. Clinicians will use the Eko CORE and/or Eko CORE 500 device(s) in real clinical settings to collect normal and abnormal lung sounds, as part of standard of care clinical practice, which will then be used to explore an ML algorithm for classifiers for wheeze, coarse crackle, fine crackle, rhonchus, stridor, rales, and cough, as well as determine any correspondences between the type and/or location of adventitious lung sounds and the type of pulmonary conditions as reported by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or diagnosed lower respiratory condition OR Presence of wheeze, coarse crackle, fine crackle, rhonchus, stridor, rales, and cough discovered during routine auscultation
* Normal patients with no adventitious lung sounds
* Adults and pediatric patients (as available)

Exclusion Criteria:

* Unable to have multiple recordings taken on chest and back (e.g. compromised mobility)
* On mechanical ventilation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects with complaints of shortness of breath or relevant diagnoses like COPD/heart failure/asthma will be screened for eligibility from the upcoming clinic schedule and then recruited during their clinical appointment. Inpatients may also be identified from the EHR and recruited from inpatient units. In order to achieve the harder-to-fill buckets, it may be necessary to directly target existing registries or patient databases, and/or bring patients in for a research-specific visit. Additionally, patients seen in clinic or in hospital with no known respiratory condition will be recruited and evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Through study completion, an average of 8-9 months
  The primary objective of this study is to collect normal and abnormal lung sounds of up to 750 patients per study site, by having clinicians use the Eko CORE and/or Eko CORE 500 device(s) in real clinical settings, as part of standard of care clinical practice which will then be used to explore an ML algorithm for classifiers for wheeze, coarse crackle, fine crackle, rhonchus, stridor, rales, and cough, as well as determine any correspondences between the type and/or location of adventitious lung sounds and the type of pulmonary conditions as reported by clinicians.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Florida
  - Jefferson Einstein Philadelphia Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No